CLINICAL TRIAL: NCT05875428
Title: A Phase 2, Single-arm, Multicenter Trial to Evaluate the Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Injection in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Mitoxantrone Hydrochloride Liposome Injection in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-033
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): The eligible patients will receive mitoxantrone hydrochloride liposome injection (20 mg/m^2) once every 4 weeks for a maximum of 8 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — Be given intravenously at 20 mg/m^2 on days 1 of each treatment cycle.

SUMMARY:
A multicenter, single-arm, phase 2 study of mitoxantrone hydrochloride liposome injection in patients with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is a phase 2, single-arm, multicenter trial to evaluate the efficacy and safety of mitoxantrone hydrochloride liposome injection in patients with R/R DLBCL. The eligible patients will receive mitoxantrone hydrochloride liposome injection (20 mg/m^2) once every 4 weeks for a maximum of 8 cycles. Patients will receive treatment until the completion of 8 cycles of treatment, disease progression, intolerable toxicity, death, loss to follow-up, withdrawal (patient's decision or investigator's decision), whichever comes first. All patients will have post-treatment follow-up for disease status until disease progression/recurrence, initiation of new antitumor therapy, or being lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study, and voluntarily sign informed consent.
2. Age ≥ 18 years old.
3. Previously treated, pathologically confirmed primary DLBCL, or DLBCL transformed from previously diagnosed indolent lymphoma (e.g., follicular lymphoma).
4. Patients are not suitable for high-dose chemotherapy combined with autologous stem cell transplantation as rescue therapy.
5. Relapsed or refractory disease after at least (≥) 2 lines of systemic therapy (including at least a regimen of anti-CD20 immunotherapy combined with cytotoxic drugs was included), there is no suitable and conventional therapy.
6. Patients have at least one measurable lesion in accordance with the Lugano evaluation criteria (version 2014):(if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progression after radiotherapy).
7. Confirmation of no objective response from the most recent therapy (at least 2 cycles of administration, and efficacy assessed as stable disease or progressive disease) or disease progression after therapy.
8. Patients must agree to provide the most recent tumor tissue section or have a biopsy of tumor tissue.
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
10. Estimated life expectancy ≥ 3 months.
11. Patients should meet the following requirements and have not received infusion of cell growth factor, blood transfusion, or blood product within 14 days of the hematology test:

    1. Absolute value of neutrophils ≥ 1.5 × 10^9/L; Hemoglobin≥80g/L; Platelet ≥ 75 × 10^9/L;
    2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; AST and ALT ≤ 5 × ULN for patients with liver metastasis. Total bilirubin ≤1.5 × ULN (≤ 3 × ULN for patients with Gilbert syndrome).
    3. Creatinine clearance ≥ 50 mL/min or serum creatinine ≤ 1.5 × ULN。
    4. Coagulation function: prothrombin time or activated partial thromboplastin time≤ 1.5 × ULN, and international normalized ratio ≤ 1.5.
12. Female patients of childbearing age must have a negative pregnancy test at the time of enrollment within one week, and must agree to use an effective method of contraception from the study initiation until at least 4 months after the last treatment; Male patients must agree to use an effective method of contraception from the study initiation until at least 6 months after the last treatment. During the study, oocyte donation of female patients and sperm donation of male patients are not allowed.
13. COVID-19 patients without related symptoms after two weeks can be enrolled.

Exclusion Criteria:

1. Primary central nervous system lymphoma, unclassified B-cell lymphoma between DLBCL and classical Hodgkin's lymphoma, primary effusion lymphoma, plasmablastic lymphoma or DLBCL transformed from previously diagnosed non-indolent lymphoma.
2. Patients with active central nervous system and meninx involvement.
3. Previously treated with mitoxantrone or mitoxantrone liposome.
4. Previously treated with adriamycin or other anthracyclines, with the total cumulative dose (doxorubicin equivalent) > 400 mg/m^2.
5. Previously treated with chimeric antigen receptor T-cell.
6. History of autologous hematopoietic stem cell transplantation or allogeneic hematopoietic stem cell transplantation within 6 months prior to screening.
7. Patients With interstitial lung disease that requires treatment.
8. History of other malignant tumor within 5 years, except for DLBCL in this trial or resected locally cancer that has been cured (e.g.basal cell or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
9. Participating in any other intervention clinical trials within 4 weeks prior to the first dose except for participation in an observational (non-interventional) clinical study or the follow-up phase of an interventional study.
10. Any steroid hormone treatment within 4 weeks prior to the first dose, chemotherapy and targeted therapy within 28 days, radiotherapy within 14 days, antibody therapy within 28 days, Chinese herbal treatment within 14 days.
11. Adverse events from the previous treatment have not resolved to ≤ Grade 1 (except for alopecia, hyperpigmentation).
12. HIV infection, active hepatitis B (positive for HBsAg, or positive for HBcAb with positive for HBV-DNA PCR), active hepatitis C(positive for anti-HCV with positive for HCV-RNA PCR), or active syphilis infection; for patients with HBV infection, consider enrolment if the disease is under control.
13. Patients with active pulmonary tuberculosis.
14. Any active infections requiring systemic or venous anti-infective treatment.
15. Patients with major surgery within 4 weeks prior to the first dose, and not recovered from any previous creative operation.
16. Any of the following conditions occurs in cardiac function:

    1. Electrocardiographic examination: QTc >480 msec;
    2. Clinically significant arrhythmias, including but not limited to complete left bundle branch block or Second-degree atrioventricular block disease, PR> 250 msec;
    3. Any risk that increase prolonged QTc or arrhythmia events, for example uncorrectable hypokalemia, hereditary long QT syndrome, and patients treated with medications that prolong QT intervals but discontinuation for less than 15 days;
    4. History of congestive heart failure, New York Heart Association (NYHA)≥grade 2;
    5. The cardiac ejection fraction is less than 50% or lower than the lower limit of the laboratory test value range of the research center;
    6. History of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, history of clinically significant pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months prior to the first dose.
17. History of allergy and contraindications to the same class and excipients of the experimental drug.
18. Pregnant or breastfeeding women;
19. Not suitable for this study as determined by the investigator due to other reasons (e.g.uncontrolled hypertension, uncontrolled diabetes, active bleeding, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by the IRC | Throughout the study period, up to approximately 2 years
  ORR (objective response rate) assessed by the Independent Review Committee (IRC)

SECONDARY OUTCOMES:
ORR assessed by investigators | Throughout the study period, up to approximately 2 years
  ORR (objective response rate) assessed by investigators
DCR | Throughout the study period, up to approximately 2 years
  Disease control rate
DOR | Throughout the study period, up to approximately 2 years
  Duration of response
PFS | Throughout the study period, up to approximately 2 years
  Progression-free survival
OS | Throughout the study period, up to approximately 2 years
  Overall survival
TEAE | Throughout the study period, up to approximately 2 years
  Treatment emergent adverse event
Blood concentrations of total and free mitoxantrone | Throughout the study period, up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No